CLINICAL TRIAL: NCT01847573
Title: A Phase 1b Open Label, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of HT-100 in Patients With Duchenne Muscular Dystrophy
Brief Title: Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses of HT-100 in Duchenne Muscular Dystrophy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Dosing stopped
Sponsor: Processa Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HALO-DMD-01; HALO (Other: Akashi Therapeutics)
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2019-03

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: halofuginone hydrobromide; anti-fibrotic; anti-inflammatory; muscle regeneration; protein synthesis inhibitor
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1: HT-100 tablet, Dose 1 (Experimental): * Single dose administration: Dose 1
  * Multiple dose administration: Dose 1
  Interventions: Drug: HT-100
- Cohort 2: HT-100 tablet, Dose 2 (Experimental): * Single dose administration: Dose 2
  * Multiple dose administration: Dose 2
  Interventions: Drug: HT-100
- Cohort 3: HT-100 tablet, Dose 3 (Experimental): * Single dose administration: Dose 3
  * Multiple dose administration: Dose 3
  Interventions: Drug: HT-100
- Cohort 4a: HT-100 tablet, Dose 4 (Experimental): * Single dose administration: Dose 4
  * Multiple dose administration: Dose 4
  Interventions: Drug: HT-100
- Cohort 4b: HT-100 tablet, Dose 5 (Experimental): * Multiple dose administration: Dose 5
  Interventions: Drug: HT-100
- Cohort 5: HT-100 tablet, Dose 6 (Experimental): * Multiple dose administration: Dose 5
  Interventions: Drug: HT-100

INTERVENTIONS:
Drug: HT-100 — May be administered in either fed or fasted state
  Other Names: halofuginone hydrobromide delayed-release tablet

SUMMARY:
The main purpose of this study is to test the safety and tolerability of different, increasing doses of an experimental medication called HT-100 in boys and young men with Duchenne muscular dystrophy (DMD). The study medication, HT-100, is a medicine that may help promote healthy muscle regeneration, diminish inflammation and the resulting damage to muscle, and decrease the scar tissue that forms in the muscles of children with DMD. In this study, pharmacokinetic sampling, or measurements of the amount of HT-100 in the bloodstream will also be taken.

ELIGIBILITY:
Main Inclusion Criteria:

* Ambulatory or non-ambulatory
* Diagnosis of DMD with confirmation of minimal to no dystrophin
* Corticosteroid naive or on therapy for at least 12 months (stable dose and regimen)

Main Exclusion Criteria:

* Recent, substantial change in use of cardiac medications or medications affecting muscle function
* Inability to undergo magnetic resonance imaging (MRI)
* Significantly compromised cardio-respiratory function
* Prior treatment with another investigational product in past 6 months

Ages: 6 Years to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2013-05; Primary Completion 2016-03-30 (Actual); Study Completion 2016-03-30 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of administering single and multiple ascending doses of HT-100 in DMD boys | 1 week
  Safety profile by review of adverse events (AEs), physical examination findings, clinical laboratory test results, and other diagnostic testing

SECONDARY OUTCOMES:
Pharmacokinetic plasma profile of halofuginone after single and multiple dose administration of HT-100 in DMD boys | 1 week
  Halofuginone plasma concentrations
Safety and tolerability of administering multiple ascending doses of HT-100 in DMD boys over 4 weeks | 4 weeks
  Safety profile by review of AEs, physical examination findings, clinical laboratory test results, and other diagnostic testing
Early pharmacodynamic signals of HT-100 after 4 weeks of continuous dosing in DMD boys | 4 weeks
  Pharmacodynamic measures relevant to DMD pathology:
  * Pulmonary function
  * Motor function
  * Muscle composition
  * Biochemical and imaging markers

CONTACTS AND LOCATIONS:
Overall Officials: Diana M Escolar, MD, Study Director — Akashi Therapeutics
Locations (5):
- United States (5):
  - University of California, Davis Medical Center, Sacramento, California
  - Kennedy Krieger Institute, Johns Hopkins School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio

REFERENCES:
- See also: Sponsor company website — http://www.akashirx.com/